CLINICAL TRIAL: NCT05254860
Title: Continuous Locked Non-barbed Suture for Mesh Fixation During Laparoscopic Ventral Rectopexy for Severe Rectal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Principal Investigator, Andrea Morciano, Principal Investigator, Azienda Ospedaliera Cardinale G. Panico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901Gineco
Record Dates: First submitted 2022-02-13; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Rectal Prolapse
Keywords: ventral rectopexy; laparoscopy; prolapse
MeSH Terms: conditions — Rectal Prolapse; Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interrupted suture (Experimental)
  Interventions: Procedure: LPS Ventral Rectopexy
- Continous suture (Experimental)
  Interventions: Procedure: LPS Ventral Rectopexy

INTERVENTIONS:
Procedure: LPS Ventral Rectopexy — Continuous Locked Suture vs Traditional 6-points suture for Laparoscopic Ventral Rectopexy to verify if the operative time of a standard laparoscopic ventral rectopexy for the treatment of severe rectal prolapse could be further reduced using continuous locked suture vs traditional 6-points suture for mesh fixation

SUMMARY:
This prospective randomized pilot study is aimed to verify if the operative time of a standard laparoscopic ventral rectopexy for the treatment of severe rectal prolapse could be further reduced using a continuous locked suture vs. conventional single 6-points suture for mesh fixation.

DETAILED DESCRIPTION:
Introduction Laparoscopic ventral rectopexy could be considered the gold standard procedure for rectal prolapse because provides the potential to combine the success rates of an abdominal approach with the faster recovery associated with a minimally invasive technique. Tissue dissection and mesh placement may also be facilitated by the magnification and field of view permitted by the laparoscopic approach. These benefits must be balanced against a longer operating time from 150 to 250 minutes according to surgeons' experience. This prospective randomized pilot study is aimed to verify if the operative time of a standard laparoscopic ventral rectopexy for the treatment of rectal prolapse could be further reduced using using a continuous locked suture vs. conventional 6-points single suture for mesh fixation.

Secondary endopoints of this comparison are incidence of intra- or postoperative complications estimated blood loss, postoperative pain (evaluated by VAS), days of hospitalization and costs for the health care system.

Statistical Analysis and Study Design This is a single Institution prospective randomized clinical trial conducted at the Pia Fondazione Panico of Tricase, Italy.

To have an imbalanced results and to reduce any bias, a randomization list has been checked.

Probability (p) values will be considered to be statistically significant at the <0.05 level.

There will be recruited 25 patients to treat using continuous locked suture and 25 patients to treat with standard 6-points single suture for mesh fixation comparing these two techniques in terms of operative time, estimated blood loss and other intra- or post operative complications, postoperative pain, days of hospitalization, costs. All patients will be adequately informed and inserted in the study only after having read and signed an informed consent. Diagnostic, clinical and surgical data of each patient will be prospectively recorded. At the end of the procedure, a schedule will be compiled with intraoperative data. All clinical and histologic data will be recorded prospectively using a database. Pain associated with the procedure will be evaluated by a subjective assessment (analysis of VAS scale values reported by patients at 8 and 24 hours after surgery). Post-operative complications will be evaluated during the first 30 days after surgery according to Dindo's classification.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Age ≤ 80 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* Physiologic, surgical or iatrogenic menopause.
* No previous major abdominal surgical procedures For diseases
* POP-Q stage III/IV for anterior and/or apical compartment; stage <III for posterior compartment.
* No uterine cervix dysplasia or endometrial disorders.
* No uterine size larger than conform 10 weeks gestation

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Operative time | 1 year
  Operative time for RVL will be calculated from the entrance to exit from the abdominal cavity

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morciano, M.D., Principal Investigator — Pia Fondazione Panico

REFERENCES:
- [Derived] Morciano A, Caliandro D, Campagna G, Panico G, Giaquinto A, Fachechi G, Zullo MA, Tinelli A, Ercoli A, Scambia G, Cervigni M, Marzo G. Laparoscopic ventral rectopexy plus sacral colpopexy: continuous locked suture for mesh fixation. A randomized clinical trial. Arch Gynecol Obstet. 2022 Nov;306(5):1573-1579. doi: 10.1007/s00404-022-06682-2. Epub 2022 Jul 15. PMID 35835920